CLINICAL TRIAL: NCT03309046
Title: Interventions for Parent Caregivers of Injured Military/Veteran Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memphis VA Medical Center (U.S. Federal Agency)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linda O. Nichols, Ph.D., Co-Director Caregiver Center, Memphis VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14029002
Record Dates: First submitted 2017-10-05; First posted 2017-10-13 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic
Keywords: Parents; Caregivers; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REACH Individual Session (Experimental): The individual sessions intervention focuses on education, skills building, and support. It will be delivered in six sessions by telephone over three months. A Caregiver Notebook will include comprehensive materials for all sessions and topics. Treatment fidelity will be monitored and ensured through assessment of intervention delivery, receipt, and enactment. The intervention is targeted and individualized to the concerns of the specific caregiver and care recipient through a risk assessment. The Risk Assessment (RA) assesses the main caregiving risk areas for the specific caregiving dyad. The RA is used to tailor the intervention for care recipient behaviors or safety issues and/or caregiver centered issues/concerns related to health, physical and emotional well being, and/or social support.
  Interventions: Other: REACH Individual Session
- Education Webinar (Active Comparator): For the education webinar sessions, topics addressing each of the caregiving risk factors topics but without the skills building or cognitive restructuring components present in the individual intervention sessions will be available online in webinars. The education webinar sessions will focus on general information about post 9/11 concerns, problem behaviors, caregiver health, caregiver emotional well-being, and red flags. Education webinar session participants will not receive the Caregiver Notebook until they have completed their 6 month interviews. Parents will be able to view all 6 webinars at any time during the first 3 months. Each session will last approximately thirty minutes through PowerPoint slide presentation format with a pre-recorded script.
  Interventions: Other: Education Webinar

INTERVENTIONS:
Other: REACH Individual Session — Individual telephone session with parent
  Arms: REACH Individual Session
Other: Education Webinar — Videos with information on caregiving
  Arms: Education Webinar

SUMMARY:
This randomized clinical trial will test a behavioral caregiving intervention that has been used successfully for dementia and spinal cord injury caregivers to provide services to stressed and burdened parent caregivers of post 9/11 service members/veterans. This intervention is six intensive individual sessions that will teach problem solving, cognitive restructuring and stress reduction targeted to an individual assessment of the care dyad's needs. It will be compared to another method of delivering content, education webinar sessions, which are analogous to the usual standard of care and will function as an attention control arm. The objective of the study is to determine which of these delivery mechanisms is more effective at helping parent caregivers of injured post 9/11 returning troops to improve their depression, anxiety, and burden, and to determine the feasibility of using individual sessions with this population of caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. Identify as a parent who serves as the primary/main caregiver for a post 9/11 service member or veteran with a diagnosis of traumatic brain injury or post traumatic stress disorder or physical injury and at least 1 activity of daily living limitation or 2 or more instrumental of daily living limitations;
2. provide 3 hours or more of care per day for at least 6 months;
3. endorse at least 2 caregiving stress behaviors (overwhelmed, often needing to cry, angry/frustrated, cut off from family/friends, moderate/high levels of stress, and declining health); and
4. have a telephone.
5. Internet access is desirable but not mandatory.

Exclusion Criteria:

1. current diagnosis of schizophrenia or other major mental illness; or
2. auditory impairment that would make telephone use difficult

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda O Nichols, PhD, Principal Investigator — Memphis VAMC
Locations (1):
- Memphis VA Medical Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be available if requested

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | REACH Individual Session | Education Webinar
Started | 82 | 81
Completed | 78 | 64
Not Completed | 4 | 17
Not completed — Withdrawal by Subject | 4 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REACH Individual Session | Education Webinar | Total
Number analyzed (Participants) | 82 | 81 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (7.3) | 60.1 (6.3) | 60.2 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 72 | 146
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 6
  Not Hispanic or Latino | 76 | 81 | 157
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 20 | 6 | 26
  White | 59 | 70 | 129
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 82 | 81 | 163
Depression [Mean (Standard Deviation); unit: units on a scale] — Measured by PHQ-9, score ranges from 0-27. Higher scores indicate more depression. Cut points for depression are <5 (minimal), <10 (mild), <15 (moderate), <20 (moderately severe), or >20 (high/severe).
  units on a scale | 6.0 (4.3) | 7.3 (5.8) | 6.6 (5.2)
Anxiety [Mean (Standard Deviation); unit: units on a scale] — Measured by the GAD-7, score range is 0-21. Higher scores indicate more anxiety. Cut points of 5, 10, and 15 represent mild, moderate, and severe levels of anxiety.
  units on a scale | 6.6 (4.7) | 7.2 (4.6) | 6.9 (4.7)
Burden [Mean (Standard Deviation); unit: units on a scale] — Measured by the Zarit Burden Inventory, score ranges from 0-48. Higher scores indicate greater burden with > 17 indicating severe/high burden.
  units on a scale | 15.7 (8.6) | 17.9 (8.9) | 16.8 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Depression - Patient Health Questionnaire - 9 (PHQ-9)
Description: The PHQ-9 has 9 items based on the DSM-IV depression diagnostic criteria. Time Frame: All questions refer to the past two weeks. Scaling: 0 (not at all) to 3 (nearly every day). On the PHQ-9, major depressive syndrome is suggested if #1 or #2 and 5 or more items are ranked positive (at least "more than half the days," count #9 if present at all). Other Depressive Syndrome suggested if #1 or #2 and two, three, or four of #1-9 are at least "More than half the days" (count #9 if present at all).
  Score ranges from 0-27. Higher scores indicate greater depression. Scores are summed to characterize depression as minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19), or high/severe (20-27).
Time Frame: 6 months
Population: intention-to-treat, with participants analyzed according to initial arm assignments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | REACH Individual Session | Education Webinar
Number analyzed (Participants) | 82 | 81
units on a scale | 4.4 (3.4) | 6.3 (4.9)

2. Primary Outcome: Anxiety - Generalized Anxiety Disorder (GAD-7). Time Frame: All Questions Refer to the Past Two Weeks.
Description: the GAD-7 contains a 7-item checklist of symptoms of GAD. All questions refer to the past two weeks. Scaling: 0 (not at all) to 3 (nearly every day)
  # of Items: 7-items. Scaling: 0 (not at all) to 3 (nearly every day).
  Scoring for each item ranges from 0 (not at all) to 3 (nearly every day) for an overall score of 0 to 21; higher scores equal more anxiety. Several cut points have been put forward for different purposes. A cut point of 10 identifies cases of generalized anxiety disorder. Cut points of 5, 10, and 15 represent mild, moderate and severe anxiety.
Time Frame: 6 months
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | REACH Individual Session | Education Webinar
Number analyzed (Participants) | 82 | 81
units on a scale | 5.3 (4.3) | 6.8 (5.1)

3. Primary Outcome: Burden - Zarit Burden Interview (ZBI-12)
Description: # of items: 12 items Scaling: 0 (Never) to 4 (Nearly Always) Total score ranges from 0-48, Higher scores indicate greater burden with > 17 indicating severe/high burden.
Time Frame: 6 months
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | REACH Individual Session | Education Webinar
Number analyzed (Participants) | 82 | 81
units on a scale | 13.4 (8.5) | 16.1 (9.7)

ADVERSE EVENTS:
Time Frame: six months
Description: Study intervention was either talking to a Coach or watching a video
Arm/Group | REACH Individual Session | Education Webinar
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/81
Other Adverse Events (participants affected / at risk) | 0/82 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-05-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT03309046/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT03309046/ICF_001.pdf